CLINICAL TRIAL: NCT05949931
Title: A Randomized, Open, Multicenter Phase II Clinical Trial of Pianzumab Combined With AVD Regimen in the Treatment of Newly-diagnosed Advanced Classic Hodgkin Lymphoma (PENAHL Study)
Brief Title: Pianzumab Combined With AVD Regimen in the Treatment of Newly-diagnosed Advanced Classic Hodgkin Lymphoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Qingqing Cai, Chief physician, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B2023-092
Record Dates: First submitted 2023-07-10; First posted 2023-07-18 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2024-08

CONDITIONS: Classic Hodgkin Lymphoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Concurrent penpulimab and AVD (Experimental): Participants will receive Penpulimab and AVD injection at the same time for a total of 6 cycles. Cycle length = 28 days, Penpulimab and AVD will be administered on D1 and D15 of each cycle.
  Interventions: Drug: Concurrent penpulimab and AVD
- Sequential penpulimab and AVD (Experimental): Participants will receive penpulimab for 3 cycles; follewed by 6 cycles of AVD; finally, penpulimab for 3 cycles. Cycle length = 28 days, Penpulimab and AVD will be administered on D1 and D15 of each cycle.
  Interventions: Drug: Sequential penpulimab and AVD

INTERVENTIONS:
Drug: Concurrent penpulimab and AVD — Participants will receive Penpulimab and AVD injection at the same time for a total of 6 cycles. Cycle length = 28 days, Penpulimab and AVD will be administered on D1 and D15 of each cycle.
  Arms: Concurrent penpulimab and AVD
Drug: Sequential penpulimab and AVD — Participants will receive penpulimab for 3 cycles; follewed by 6 cycles of AVD; finally, penpulimab for 3 cycles. Cycle length = 28 days, Penpulimab and AVD will be administered on D1 and D15 of each cycle.
  Arms: Sequential penpulimab and AVD

SUMMARY:
This study is conducted to evaluate the safety and efficiency of Penpulimab combined with AVD in patients with newly- diagnosed advanced classic Hodgkin lymphoma.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18-70 years old (when signing the informed consent form); ECOG score: 0 or 1 point; The expected survival period exceeds 3 months;
2. classic Hodgkin lymphoma (cHL) confirmed by histopathology;
3. The subject must be advanced patient, specifically defined as Ann Arbor stage III-IV or IIB with any of the following high-risk factors: ① maximum diameter of mediastinal mass/maximum diameter of thoracic cavity>0.33; ② There are large masses with a diameter of>10cm;
4. Have not received systemic anti classic Hodgkin lymphoma treatment;
5. Measurable disease ;
6. Adequate main organs function
7. Female subjects of childbearing age should agree to use contraceptives (such as Intrauterine device, contraceptives or condoms) during the study period and within 6 months after the end of the study; The serum or urine Pregnancy test was negative within 7 days before the study was included, and must be non-lactating subjects; Male participants should agree to use contraception during the study period and within 6 months after the end of the study period.

Exclusion Criteria:

1. Nodular lymphocyte dominated Hodgkin lymphoma or gray area lymphoma;
2. Classic Hodgkin lymphoma involves the central nervous system;
3. Subjects who have or are suspected to have active autoimmune diseases within the past 2 years, or have previously suffered from autoimmune diseases and are currently at high risk of recurrence and require systemic treatment；
4. Subjects who need to use glucocorticoid (>10mg/day prednisone Equivalent dose) or other immunosuppressive drugs for systemic treatment within 14 days before the first administration.
5. Inoculate or expect to receive live or attenuated live vaccines or mRNA vaccines within 4 weeks before the first administration;
6. Received allogeneic organ transplantation or allogeneic hematopoietic stem cell transplantation;
7. Known to have active pulmonary tuberculosis;
8. Having a history of immunodeficiency, including HIV positive or suffering from other acquired or congenital immunodeficiency diseases;
9. Subjects with a known history of interstitial pneumonia, a history of non-infectious pneumonia, or highly suspected cases of interstitial pneumonia;
10. Patients with evidence of bleeding constitution or medical history; Within 4 weeks before the first medication, any ≥ CTC AE level 3 bleeding events (such as digestive tract bleeding, perforation, etc.) occur;
11. Concomitant diseases and medical history:

    1. Has experienced or currently suffers from other malignant tumors within 3 years.
    2. Multiple factors affecting oral medicine (such as inability to swallow, chronic diarrhea and Bowel obstruction);
    3. Patients with a history of abuse of psychotropic substances who are unable to quit or have mental disorders;
    4. Subjects with any severe and/or uncontrollable disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Complete response rate （CRR） | From first injection to 24 weeks (Arm 1) From first injection to 48 weeks (Arm 2)
  Percentage of participants achieving complete response evaluated by the Independent Review Committee (IRC) at the end of all treatment courses

SECONDARY OUTCOMES:
Complete response rate （CRR） | From first injection to 24 weeks (Arm 1) From first injection to 48 weeks (Arm 2)
  Percentage of participants achieving complete response evaluated by researchers
Objective response rate（ORR） | From first injection to 24 weeks (Arm 1) From first injection to 48 weeks (Arm 2)
  Percentage of participants achieve complete response and partial response
Progression-free Survival (PFS) | Up to 5 years
  From randomization to the first occurrence of disease progression as determined by the investigator, or death due to any cause, whichever occurs first
Overall survival (OS) | Up to 5 years
  From randomization to the time of death from any cause.
Safety indicators | Up to 5 years
  The incedence of all adverse events (AEs), serious adverse events (SAEs) and treatment-related adverse events (TEAEs).

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen Universitiy Cancer Center, Sun Yat-Sen University, Guangzhou, Guangdong, China